CLINICAL TRIAL: NCT01443494
Title: High Mean Arterial Pressure Target Improves Microcirculation in Septic Shock Patients With Previous Hypertension
Brief Title: High MAP in Septic Shock With Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Jingyuan,Xu, ZhongDa Hospital, Southeast University, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SoutheastUChina2011ZDllKY03.0
Record Dates: First submitted 2011-09-28; First posted 2011-09-29 (Estimated); Results first posted 2014-06-16 (Estimated); Last update posted 2017-07-06 (Actual); Status verified 2017-06

CONDITIONS: Septic Shock
Keywords: septic shock; microcirculation; norepinephrine; fluid
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NE group (Experimental): Adjust NE dose to titrate MAP to usual level regardless of fluid responsiveness when after EGDT.
  Interventions: Other: NE

INTERVENTIONS:
Other: NE — norepinephine

SUMMARY:
We hypothesized that the increase in MAP from 65 mmHg to patients' usual level improved sublingual microcirculation.

DETAILED DESCRIPTION:
The effect of mean arterial pressure (MAP) titration to higher level on microcirculation in septic shock patients with previous hypertension remains unknown. Our goal was to assess the effect of MAP titration to patients' usual level on microcirculation in septic shock patients with previous hypertension. We hypothesized that the increase in MAP from 65 mmHg to patients' usual level improved sublingual microcirculation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with septic shock for less than 24 hours
* Fluid resuscitation was performed according to the guideline for treating septic shock to maintain the central venous pressure (CVP) for more than 8 mm Hg and central venous oxygen saturation for more than 70%
* Patients requiring norepinephrine (NE) to maintain a MAP of 65 mm Hg. Septic shock patients with fluid resuscitation after CVP > 8mmHg and mean blood pressure > 65 mmHg

Exclusion Criteria:

* Pregnancy
* Age < 18 years
* Inability to acquire the usual level of MAP
* Refusal of consent by the patient or relative
* Participation in other trials during the last three months
* Hypertensive patients without hypertension treatment

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Haibo Qiu, MD,PhD, Study Director — Southeast University
Locations (1):
- Zhongda Hospital Southeast University, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Sakr Y, Dubois MJ, De Backer D, Creteur J, Vincent JL. Persistent microcirculatory alterations are associated with organ failure and death in patients with septic shock. Crit Care Med. 2004 Sep;32(9):1825-31. doi: 10.1097/01.ccm.0000138558.16257.3f. PMID 15343008
- [Background] Correa TD, Vuda M, Takala J, Djafarzadeh S, Silva E, Jakob SM. Increasing mean arterial blood pressure in sepsis: effects on fluid balance, vasopressor load and renal function. Crit Care. 2013 Jan 30;17(1):R21. doi: 10.1186/cc12495. PMID 23363690
- [Background] Beloncle F, Lerolle N, Radermacher P, Asfar P. Target blood pressure in sepsis: between a rock and a hard place. Crit Care. 2013 Mar 26;17(2):126. doi: 10.1186/cc12543. PMID 23534963
- [Background] Sevransky JE, Nour S, Susla GM, Needham DM, Hollenberg S, Pronovost P. Hemodynamic goals in randomized clinical trials in patients with sepsis: a systematic review of the literature. Crit Care. 2007;11(3):R67. doi: 10.1186/cc5948. PMID 17584921
- [Background] LeDoux D, Astiz ME, Carpati CM, Rackow EC. Effects of perfusion pressure on tissue perfusion in septic shock. Crit Care Med. 2000 Aug;28(8):2729-32. doi: 10.1097/00003246-200008000-00007. PMID 10966242
- [Background] Jhanji S, Stirling S, Patel N, Hinds CJ, Pearse RM. The effect of increasing doses of norepinephrine on tissue oxygenation and microvascular flow in patients with septic shock. Crit Care Med. 2009 Jun;37(6):1961-6. doi: 10.1097/CCM.0b013e3181a00a1c. PMID 19384212
- [Background] Dubin A, Pozo MO, Casabella CA, Palizas F Jr, Murias G, Moseinco MC, Kanoore Edul VS, Palizas F, Estenssoro E, Ince C. Increasing arterial blood pressure with norepinephrine does not improve microcirculatory blood flow: a prospective study. Crit Care. 2009;13(3):R92. doi: 10.1186/cc7922. Epub 2009 Jun 17. PMID 19534818
- [Background] Thooft A, Favory R, Salgado DR, Taccone FS, Donadello K, De Backer D, Creteur J, Vincent JL. Effects of changes in arterial pressure on organ perfusion during septic shock. Crit Care. 2011;15(5):R222. doi: 10.1186/cc10462. Epub 2011 Sep 21. PMID 21936903
- [Derived] Xu JY, Ma SQ, Pan C, He HL, Cai SX, Hu SL, Liu AR, Liu L, Huang YZ, Guo FM, Yang Y, Qiu HB. A high mean arterial pressure target is associated with improved microcirculation in septic shock patients with previous hypertension: a prospective open label study. Crit Care. 2015 Mar 30;19(1):130. doi: 10.1186/s13054-015-0866-0. PMID 25887027

RESULTS

PARTICIPANT FLOW:
Groups:
- Septic Shock Patients Despite EGDT With Hypertension: Patients with previous hypertension requiring norepinephrine to maintain a MAP of 65 mm Hg despite fluid resuscitation to central venous pressure above 8 mm Hg.
Period: Overall Study
Arm/Group | Septic Shock Patients Despite EGDT With Hypertension
Started | 19
Completed | 19
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Detailed enquiry about the target MAP to their next kin was performed in all of the patients.
Arm/Group | Septic Shock Patients Despite EGDT With Hypertension
Number analyzed (Participants) | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 13
Region of Enrollment [Number; unit: participants]
  China | 19

OUTCOME MEASURES:

1. Primary Outcome: Mean Arterial Pressure
Description: As chronic hypertensive patients were supposed to have undergone more blood pressure measurements in daily life than non-hypertensive ones, the averaged MAP acquired from patients' physical examination records of the last two years was registered and assumed as patients' usual level of MAP and target MAP. If patients' medical records were incomplete, a detailed enquiry about the target MAP to their next kin was performed.
  After stabilization for 30 min, basal measurements including hemodynamic and microcirculatory measurements were taken, 20 min apart, the NE doses were increased to titrate MAP to the target level. Patients were allowed to stabilize for 30 min before taking new measurements.
Time Frame: Target MAP stabilization for 30 min
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Septic Shock Patients Despite EGDT: After stabilization for 30 min, basal measurements including hemodynamic and microcirculatory measurements were taken, 20 min apart, the NE doses were increased to titrate MAP to the target level. Patients were allowed to stabilize for 30 min before taking new measurements.
Arm/Group | Septic Shock Patients Despite EGDT
Number analyzed (Participants) | 19
mmHg | 90 (7)

2. Secondary Outcome: Perfused Vessel Density
Description: Increasing MAP from 65 mm Hg to target level. The sublingual microcirculation was measured by sidestream dark field, including the parameters of perfused vessel density
Time Frame: Target MAP stabilization for 30 min
Measure: Mean (Standard Deviation); unit: vessels/mm^2
Arm/Group | Septic Shock Patients Despite EGDT
Number analyzed (Participants) | 19
vessels/mm^2 | 12.08 (2.52)

ADVERSE EVENTS:
Time Frame: During the study procedure for about 2 hours
Groups:
- Septic Shock Patients Despite EGDT: Patients requiring norepinephrine to maintain a MAP of 65 mm Hg despite fluid resuscitation to central venous pressure above 8 mm Hg.
Arm/Group | Septic Shock Patients Despite EGDT
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 0/19

LIMITATIONS AND CAVEATS:
Firstly, cardiac output was monitored by NICOM system to minimize the invasive operation.

Secondly, the number of patients enrolled in the study was relatively small. Next, immediate changes of the increase in MAP were investigated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes